CLINICAL TRIAL: NCT04152603
Title: Better Research Interactions for Every Family
Acronym: BRIEF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: University of Washington (Other); National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Stephanie Kraft, Assistant Professor, Seattle Children's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: K01HG010361 (NIH); K23HD103872 (NIH)
Record Dates: First submitted 2019-10-31; First posted 2019-11-05 (Actual); Results first posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Respect; Trust; Study Enrollment

STUDY DESIGN:
Intervention Model Description: The BRIEF Educational Module for research recruitment team members is intended to teach evidence-based approaches to improving participant experiences with research recruitment. It has three components: (1) asynchronous pre-work, including multimedia materials and an individual worksheet (approx. 30 min); (2) one synchronous in-person (or virtual if necessary) session, including didactics, discussions, and practice scenarios (approx. 90 min); and (3) an asynchronous, individual follow-up phone call to review individual questions (approx. 15 min).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): Enrollment rates, parent/LAR-reported trust in research, and parent/LAR-reported experiences of respect during research recruitment before implementation of the BRIEF intervention.
- BRIEF Arm (Experimental): Enrollment rates, parent/LAR-reported trust in research, and parent/LAR-reported experiences of respect during research recruitment after implementation of the BRIEF intervention.
  Interventions: Behavioral: BRIEF Educational Module

INTERVENTIONS:
Behavioral: BRIEF Educational Module — The BRIEF Educational Module for research recruitment team members is intended to teach evidence-based approaches to improving participant experiences with research recruitment. It has three components: (1) asynchronous pre-work, including multimedia materials and an individual worksheet (approx. 30 min); (2) one synchronous in-person (or virtual if necessary) session, including didactics, discussions, and practice scenarios (approx. 90 min); and (3) an asynchronous, individual follow-up phone call to review individual questions (approx. 15 min).
  Arms: BRIEF Arm

SUMMARY:
This is a study of the feasibility of implementing a modified recruitment approach, the Better Research Interactions for Every Family (BRIEF) Intervention, within a neonatal clinical trial. This intervention has two distinct aims: 1) improve the experience for parents asked to enroll their infant in a neonatal clinical trial; and 2) decrease disparities in enrollment within a neonatal clinical trial. The investigators will apply the BRIEF within a single site neonatal RCT, the Darbe plus IV Iron (DIVI) study, using a pre/post approach. The intervention will be implemented approximately halfway through recruitment for the DIVI study. The objectives of this study are to assess feasibility, gain preliminary experience to drive further refinement, and provide effect estimates for a future RCT of the BRIEF intervention.

DETAILED DESCRIPTION:
The BRIEF Intervention will test the hypothesis that an evidence-based, researcher-facing educational module will improve the enrollment process for eligible families and increase diversity of populations enrolled in research. These in turn will improve the generalizability of neonatal clinical trials. The BRIEF Intervention is an educational module based on data about how research teams can approach families about research in a more equitable and respectful manner. The intervention will be implemented approximately halfway through DIVI study recruitment. The BRIEF team will measure outcomes, comparing before versus after the BRIEF Intervention is implemented, across three groups of participants:

1. Neonates eligible for participation in the DIVI study, identified through the records of the DIVI team. Research activities for this group are limited to extraction of targeted demographic and clinical data from the medical record by the BRIEF study team.
2. Parents/legally authorized representatives (LARs) of infants approached for the DIVI study who will be invited to take a survey about their experience being approached for the DIVI study, including questions about perceived respect and a validated scale to measure trust in medical researchers. Those who enroll in DIVI as well as those who decline to enroll in DIVI will be eligible to take the survey. The survey will also give them an opportunity to opt in to potentially be contacted for an interview, in which they will be asked open-ended questions about their experience being approached for the DIVI study.
3. DIVI study team members involved in recruitment. At or near the start of the DIVI study, the BRIEF team will obtain a list of contact information for each member of the DIVI team who will be involved in recruitment. The BRIEF team will contact each person individually to review and sign the BRIEF study consent form. The DIVI team will be asked to participate in the BRIEF educational module, which includes asynchronous and synchronous components, complete brief self-assessments of their consent discussions with families both before and after the intervention, and audio-record a subset of DIVI consent discussions so that the BRIEF team can assess fidelity to intervention components.

ELIGIBILITY:
Inclusion Criteria:

* Neonates (born between 24-0 and 31-6 weeks of gestation) at the University of Washington Medical Center (UWMC) eligible for inclusion in the Darbe plus IV Iron (DIVI) study; OR
* Parents or legally authorized representatives (LARs) of neonates approached for participation in the DIVI study; OR
* Members of the DIVI research team involved in recruitment.

Exclusion Criteria:

* None

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie A Kraft, JD, Principal Investigator — Seattle Children's Hospital; Elliott M Weiss, MD, MSME, Principal Investigator — Seattle Children's Hospital
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started on October 10, 2022 and ended on December 31, 2023. All recruitment took place remotely.
Pre-assignment Details: Given the pre-post design of the study, participants were not pre-assigned to the control or BRIEF arm. Rather, assignment was based on the date of a participant's enrollment. Participants excluded from the study are limited to those not eligible for the partner clinical trial (DIVI study).
Groups:
- DIVI Study Team: Group consists of the partner study team members who received the BRIEF training.
  BRIEF Educational Module: The BRIEF Educational Module for research recruitment team members is intended to teach evidence-based approaches to improving participant experiences with research recruitment. It has three components: (1) asynchronous pre-work, including multimedia materials and an individual worksheet (approx. 30 min); (2) one synchronous in-person (or virtual if necessary) session, including didactics, discussions, and practice scenarios (approx. 90 min); and (3) an asynchronous, individual follow-up phone call to review individual questions (approx. 15 min).
Period: Overall Study
Arm/Group | Control Arm | BRIEF Arm | DIVI Study Team
Started | 52 | 77 | 9
Neonates | 33 | 56 | 0
Parents/LARs | 19 | 21 | 0
Completed | 52 | 77 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm | BRIEF Arm | DIVI Study Team | Total
Number analyzed (Participants) | 52 | 77 | 9 | 138
Age, Continuous [Mean (Full Range); unit: Years] — Population: Each row represents a subset of the overall population. Neonate age data not collected and analyzed.
  Years
    Neonates: number analyzed (Participants) | 0 | 0 | 0 | 0
    Parents/LARs: number analyzed (Participants) | 19 | 21 | 0 | 40
    Parents/LARs | 31 [20 to 42] | 34 [23 to 43] |  | 32 [20 to 43]
    DIVI Team: number analyzed (Participants) | 0 | 0 | 9 | 9
    DIVI Team |  |  | 44 [26 to 73] | 44 [26 to 73]
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Each row represents a subset of the overall population.
  Participants
    Neonates: number analyzed (Participants) | 33 | 56 | 0 | 89
    Neonates: Female | 15 | 19 |  | 34
    Neonates: Male | 18 | 31 |  | 49
    Neonates: Unknown | 0 | 6 |  | 6
    Parents/LARs: number analyzed (Participants) | 19 | 21 | 0 | 40
    Parents/LARs: Female | 11 | 15 |  | 26
    Parents/LARs: Male | 8 | 5 |  | 13
    Parents/LARs: Unknown | 0 | 1 |  | 1
    DIVI Team: number analyzed (Participants) | 0 | 0 | 9 | 9
    DIVI Team: Female |  |  | 5 | 5
    DIVI Team: Male |  |  | 3 | 3
    DIVI Team: Unknown |  |  | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Each row represents a subset of the overall population.
  Participants
    Neonates: number analyzed (Participants) | 33 | 56 | 0 | 89
    Neonates: Hispanic or Latino | 5 | 13 |  | 18
    Neonates: Not Hispanic or Latino | 27 | 34 |  | 61
    Neonates: Unknown or Not Reported | 1 | 9 |  | 10
    Parents/LARs: number analyzed (Participants) | 19 | 21 | 0 | 40
    Parents/LARs: Hispanic or Latino | 7 | 7 |  | 14
    Parents/LARs: Not Hispanic or Latino | 12 | 13 |  | 25
    Parents/LARs: Unknown or Not Reported | 0 | 1 |  | 1
    DIVI Team: number analyzed (Participants) | 0 | 0 | 9 | 9
    DIVI Team: Hispanic or Latino |  |  | 1 | 1
    DIVI Team: Not Hispanic or Latino |  |  | 8 | 8
    DIVI Team: Unknown or Not Reported |  |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Each row represents a subset of the overall population.
  Participants
    Neonates: number analyzed (Participants) | 33 | 56 | 0 | 89
    Neonates: American Indian or Alaska Native | 1 | 4 |  | 5
    Neonates: Asian | 0 | 7 |  | 7
    Neonates: Native Hawaiian or Other Pacific Islander | 1 | 0 |  | 1
    Neonates: Black or African American | 6 | 12 |  | 18
    Neonates: White | 24 | 20 |  | 44
    Neonates: More than one race | 1 | 1 |  | 2
    Neonates: Unknown or Not Reported | 0 | 12 |  | 12
    Parents/LARs: number analyzed (Participants) | 19 | 21 | 0 | 40
    Parents/LARs: American Indian or Alaska Native | 0 | 1 |  | 1
    Parents/LARs: Asian | 0 | 1 |  | 1
    Parents/LARs: Native Hawaiian or Other Pacific Islander | 1 | 0 |  | 1
    Parents/LARs: Black or African American | 1 | 2 |  | 3
    Parents/LARs: White | 16 | 11 |  | 27
    Parents/LARs: More than one race | 1 | 1 |  | 2
    Parents/LARs: Unknown or Not Reported | 0 | 5 |  | 5
    DIVI Team: number analyzed (Participants) | 0 | 0 | 9 | 9
    DIVI Team: American Indian or Alaska Native |  |  | 0 | 0
    DIVI Team: Asian |  |  | 0 | 0
    DIVI Team: Native Hawaiian or Other Pacific Islander |  |  | 0 | 0
    DIVI Team: Black or African American |  |  | 1 | 1
    DIVI Team: White |  |  | 8 | 8
    DIVI Team: More than one race |  |  | 0 | 0
    DIVI Team: Unknown or Not Reported |  |  | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Study Enrollment Rates
Description: The BRIEF team will compare DIVI enrollment rates for the Neonate group before vs. after implementation of the BRIEF intervention.
Time Frame: Control Arm was assessed from baseline to the date of the intervention (pre-intervention) and the BRIEF Arm was assessed post-intervention to study completion (post-intervention), estimated at 14 months total (October 2022-December 2023).
Population: Number of BRIEF participants across the Control and BRIEF arms that either enrolled in the DIVI study or did not enroll in the DIVI study (neonates only).
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | BRIEF Arm
Number analyzed (Participants) | 33 | 56
Participants
  Enrolled in DIVI | 13 | 24
  Not Enrolled in DIVI | 20 | 32

2. Primary Outcome: Patient Trust in Research
Description: The BRIEF team will compare parent/LAR-reported trust in research before vs. after implementation of the BRIEF intervention, using the validated 4-Item Trust in Medical Researchers scale described in Hall et al. 2008. Each item is scored on a 1-5 scale for a maximum score of 20 and a minimum score of 4, with higher scores indicating more trust. Scores are then indexed to a scale of 0-100, again with a higher rating indicating greater levels of trust.
Time Frame: Control Arm was assessed at baseline (pre-intervention) and the BRIEF Arm was assessed at study completion (post-intervention), estimated at 14 months (October 2022-December 2023).
Population: Parents/LARs only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Arm | BRIEF Arm
Number analyzed (Participants) | 19 | 21
score on a scale | 78 (18) | 77 (11)

3. Primary Outcome: Change in Patient Experiences of Respect During Research Recruitment
Description: The BRIEF team will compare parent/LAR-reported experiences of being treated with respect during research recruitment before vs. after implementation of the BRIEF intervention. There is no relevant validated measure so this outcome will be measured using team-developed survey questions. Questions are measured on a Likert Scale, each item is scored on a 1-5 scale , with higher scores indicating greater perception of respect.
Time Frame: as for outcome 2
Population: Parents/LARs only.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Control Arm | BRIEF Arm
Number analyzed (Participants) | 19 | 21
score on a scale | 4.36 [2 to 5] | 4.76 [4 to 5]

ADVERSE EVENTS:
Time Frame: 1 year
Description: AEs are identified by self-report from study participants to the research team. SAEs and specific procedure-associated AEs are reported to the sponsor and IRB within 24 hours. In addition, all AEs are reported according to the University of Washington IRB AE reporting guidelines.
  Adverse events data were not collected from Neonates as that component of our study was limited to secondary data collection.
Groups:
- Control Arm: Enrollment rates, parent/LAR-reported trust in research, and parent/LAR-reported experiences of respect during research recruitment before implementation of the BRIEF intervention.
  Adverse events data were not collected from Neonates as that component of our study was limited to secondary data collection.
- BRIEF Arm: Enrollment rates, parent/LAR-reported trust in research, and parent/LAR-reported experiences of respect during research recruitment after implementation of the BRIEF intervention.
  BRIEF Educational Module: The BRIEF Educational Module for research recruitment team members is intended to teach evidence-based approaches to improving participant experiences with research recruitment. It has three components: (1) asynchronous pre-work, including multimedia materials and an individual worksheet (approx. 30 min); (2) one synchronous in-person (or virtual if necessary) session, including didactics, discussions, and practice scenarios (approx. 90 min); and (3) an asynchronous, individual follow-up phone call to review individual questions (approx. 15 min).
  Adverse events data were not collected from Neonates as that component of our study was limited to secondary data collection.
Arm/Group | Control Arm | BRIEF Arm
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/30
Other Adverse Events (participants affected / at risk) | 0/28 | 0/30

LIMITATIONS AND CAVEATS:
Due to limitations experienced by the partner clinical trial, we were unable to meet our desired recruitment goals for Spanish-speaking participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (5):
  • Study Protocol (2023-01-23): https://cdn.clinicaltrials.gov/large-docs/03/NCT04152603/Prot_003.pdf
  • Statistical Analysis Plan (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT04152603/SAP_004.pdf
  • Informed Consent Form: BRIEF Parent Survey (2022-05-19): https://cdn.clinicaltrials.gov/large-docs/03/NCT04152603/ICF_000.pdf
  • Informed Consent Form: BRIEF Parent Interview (2022-07-07): https://cdn.clinicaltrials.gov/large-docs/03/NCT04152603/ICF_001.pdf
  • Informed Consent Form: BRIEF Intervention (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/03/NCT04152603/ICF_002.pdf